CLINICAL TRIAL: NCT01024062
Title: Phase II Study of Weekly Paclitaxel (BMS-181339) in Patient With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA139-373
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; BMS 181339

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Solution, IV, 100 mg/m², weekly for 6 of 7 weeks, until disease progression or unacceptable toxicity became apparent
  Other Names: Taxol; BMS-181339

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of paclitaxel given weekly in patients with advanced or recurrent non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Patients with no prior chemotherapy who meet either of the listed below:
* Patient with stage IIIB or IV disease
* Patients with recurrent disease following potentially curative surgical resection
* Patients with previous chemotherapy up to one regimen

Exclusion Criteria:

* Patients with serious, uncontrolled medical illness
* Patients with previous therapy with taxanes

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Response rate [defined as total number of patients with complete and partial response divided by number of response-evaluable patients] based on "Response Evaluation Criteria in Solid Tumors (RECIST)" in patients with no prior chemotherapy | Each 49 day course of treatment until withdrawal or unacceptable toxicity
Safety: incidence and severity of adverse events, laboratory test abnormalities | Each 49 day course of treatment until withdrawal or unacceptable toxicity

SECONDARY OUTCOMES:
Duration of response, [measured from the time that measurement criteria are met for complete or partial response until the first date that recurrent or progressive disease is objectively documents] | Each 49 day course of treatment until withdrawal or unacceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx